CLINICAL TRIAL: NCT04578080
Title: Effect of tDCS on Motor Functions and Brain Activity in Acute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: SI284/2020
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal-tDCS & PT (Experimental): Anodal transcranial direct current stimulation (tDCS) will be applied for 20 mins before conventional physical therapy (about 1 hours). Anodal on the motor area (M1) of affected hemisphere, Cathodal on the supraorbital area of unaffected hemisphere.
  Current intensity is fixed at 1.5 mA and current will flow continuously. Physical therapist will give an intervention program base on the same basic conventional physical therapy treatment. The scope of intervention is administered to improve motor functions and brain activity.
  Interventions: Device: Transcranial direct current stimulation
- Sham-tDCS & PT (Active Comparator): Anodal transcranial direct current stimulation (tDCS) will be applied for 20 mins before conventional physical therapy (about 1 hours). Anodal on the motor area of affected hemisphere, Cathodal on the supraorbital area of affected hemisphere. Physical therapist will give an intervention program base on the same basic conventional physical therapy treatment. The scope of intervention is administered to improve motor functions and brain activity.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Anodal or Sham tDCS will be applied in 1.5 mA, 20 mins before conventional physical therapy for 5 days. All experiments will be performed in random order for each subject.

SUMMARY:
This study aims to investigate the effects of anodal tDCS combined with conventional physical therapy for 5 consecutive sessions on motor functions and brain activity in acute stroke patients at immediate and 1-month follow-up.

DETAILED DESCRIPTION:
Stroke or cerebrovascular accident is a leading cause of disabilities. Physical therapy is a standard treatment to help motor recovery after stroke. However, disabilities remained in some stroke patients despite intensive training. After stroke, there are changes of cortical excitability and brain activity in both hemispheres. Lesioned hemisphere decreases cortical excitability and increases number of low-frequency brain activity, while the non-lesioned hemisphere increases cortical excitability and increases number of high-frequency brain activity. Transcranial direct current stimulation (tDCS) is a technique which delivers weak direct current through scalp and can be used as an adjunctive treatment. Anodal tDCS can increase cortical excitability and amount of high-frequency brain activity. Increased amount of high-frequency brain activity in the lesioned hemisphere can indicate better recovery of stroke. Meta-analysis has reported the benefits of anodal tDCS for motor recovery in stroke patients. However, only few studies have investigated tDCS effects in acute phase of stroke which is a crucial time for enhancing motor recovery. This study aims to investigate the effects of anodal- and cathodal tDCS combined with conventional physical therapy for 5 consecutive sessions on motor functions and brain activity in acute stroke patients at immediate and 1-month follow-up. Participants will be randomly assigned into 2 groups (sham-, and anodal tDCS). Participants in the anodal group will receive 1.5 mA tDCS for 20 minutes before physical therapy programs for 5 consecutive sessions, while the sham group will receive sham tDCS with physical therapy. Brain activity by electroencephalography and motor performances by Fugl-Meyer Assessment and Wolf Motor Function Test will be evaluated at baseline, post-intervention (day 5), and follow-up at 1 month. We hypothesize that anodal tDCS combined with physical therapy for 5 consecutive days can immediately increase number of high-frequency brain activity and improve motor functions and this effect will last for a month compared to the sham group.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old
2. First-ever acute ischemic stroke of anterior circulation system (anterior cerebral artery or middle cerebral artery territory)
3. Stroke onset from 2-10 days
4. Having a stable medical condition
5. Alert of consciousness
6. Able to follow commands
7. Modified Rankin Scale (mRS) ≤ 4

Exclusion Criteria:

1. Hemorrhagic stroke
2. Recurrent stroke
3. Presence of other neurological disorders such as unilateral neglect
4. Presence of metal implantation, intracranial shunt, cochlear implantation or cardiac pacemakers
5. Presence of opened wound or infectious wound around scalp
6. History of epilepsy or any neurological antecedent or unstable condition which can lead to seizure
7. Body Mass Index (BMI) > 30 kg/m2
8. Received hormonal treatment
9. Ischemic heart disease and peripheral vascular ischemia
10. Last stage of kidney disease and liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Electroencephalography | 10 minutes
  Brain activity will be recorded during eyes open (5 minutes) follow by eyes close (5 minutes).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | 20 minutes
  The gold standard and widely used tool to assess sensorimotor in stroke. The item from upper limb and lower limb section will be used. The items are rated on a 3-point ordinal scale as follows: 0 = unable to perform; 1 = partial ability to perform; and 2 = near normal ability to perform.

OTHER OUTCOMES:
Wolf Motor Function Test | 5 minutes
  Two sub-items (lift a can and lift a pencil) will be evaluated in all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vimolratana O, Aneksan B, Siripornpanich V, Hiengkaew V, Prathum T, Jeungprasopsuk W, Khaokhiew T, Vachalathiti R, Klomjai W. Effects of anodal tDCS on resting state eeg power and motor function in acute stroke: a randomized controlled trial. J Neuroeng Rehabil. 2024 Jan 3;21(1):6. doi: 10.1186/s12984-023-01300-x. PMID 38172973